CLINICAL TRIAL: NCT06850051
Title: A Phase 1, Parallel, Randomized, Multi-center Study to Evaluate the Safety and Immunogenicity of Different Formulations of Multivalent Influenza and Respiratory Syncytial Virus (RSV)/Human Metapneumovirus (hMPV)/Parainfluenza Virus Type 3 (PIV3) Vaccines in Healthy Participants 18 to 49 Years of Age.
Brief Title: A Study on the Safety and Immunogenicity of Influenza, Respiratory Syncytial Virus, Human Metapneumovirus and Parainfluenza Vaccines in Adults 18 to 49 Years of Age.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VAV00030; U1111-1311-1743 (Other: WHO ICTRP)
Record Dates: First submitted 2025-02-11; First posted 2025-02-27 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Healthy Volunteers; Influenza Vaccination; Respiratory Syncytial Virus Vaccination; Parainfluenza Vaccination; Human Metapneumovirus Vaccination
Keywords: influenza; respiratory syncytial virus; parainfluenza; human metapneumovirus
MeSH Terms: conditions — Influenza, Human; Paramyxoviridae Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Group 1 trivalent influenza vaccine-hemagglutinin (TIV-HA) formulation 1 at high dose (Experimental): Participants will receive a single IM (Intramuscular) injection on day 1 of the TIV-HA vaccines according to their randomization schedule.
  Interventions: Biological: TIV-HA formulation 1 at high dose
- Group 2 TIV-HA formulation 2 at high dose (Experimental): Participants will receive a single IM (Intramuscular) injection on day 1 of the TIV-HA vaccines according to their randomization schedule.
  Interventions: Biological: TIV-HA formulation 2 at high dose
- Group 3 TIV-HA formulation 1 at low dose (Experimental): Participants will receive a single IM (Intramuscular) injection on day 1 of the TIV-HA vaccines according to their randomization schedule.
  Interventions: Biological: TIV-HA Vaccine formulation 1 at low dose
- Group 4 TIV-HA formulation 2 at low dose (Experimental): Participants will receive a single IM (Intramuscular) injection on day 1 of the TIV-HA vaccines according to their randomization schedule.
  Interventions: Biological: TIV-HA formulation 2 at low dose
- Group 5 RSV/hMPV/PIV3 formulation 1 at high dose (Experimental): Participants will receive a single IM (Intramuscular) injection on day 1 of the RSV/hMPV/PIV3 vaccines according to their randomization schedule.
  Interventions: Biological: RSV/hMPV/PIV3 formulation 1 at high dose
- Group 6 RSV/hMPV/PIV3 formulation 2 at high dose (Experimental): Participants will receive a single IM (Intramuscular) injection on day 1 of the RSV/hMPV/PIV3 vaccines according to their randomization schedule.
  Interventions: Biological: RSV/hMPV/PIV3 formulation 2 at high dose
- Group 7 RSV/hMPV/PIV3 formulation 1 at low dose (Experimental): Participants will receive a single IM (Intramuscular) injection on day 1 of the RSV/hMPV/PIV3 vaccines according to their randomization schedule.
  Interventions: Biological: RSV/hMPV/PIV3 formulation 1 at low dose
- Group 8 RSV/hMPV/PIV3 formulation 2 at low dose (Experimental): Participants will receive a single IM (Intramuscular) injection on day 1 of the RSV/hMPV/PIV3 vaccines according to their randomization schedule.
  Interventions: Biological: RSV/hMPV/PIV3 formulation 2 at low dose
- Group 9 recombinant influenza vaccine quadrivalent (RIV4) (Active Comparator): Participants will receive a single IM (Intramuscular) injection on day 1 of the RIV4 vaccine according to their randomization schedule.
  Interventions: Biological: RIV4 (Supemtek®)

INTERVENTIONS:
Biological: TIV-HA Vaccine formulation 1 at low dose — Suspension for injection in a vial. Route of administration: IM injection
  Arms: Group 3 TIV-HA formulation 1 at low dose
Biological: TIV-HA formulation 1 at high dose — Suspension for injection in a vial. Route of administration: IM injection
  Arms: Group 1 trivalent influenza vaccine-hemagglutinin (TIV-HA) formulation 1 at high dose
Biological: TIV-HA formulation 2 at low dose — Suspension for injection in a vial. Route of administration: IM injection
  Arms: Group 4 TIV-HA formulation 2 at low dose
Biological: TIV-HA formulation 2 at high dose — Suspension for injection in a vial. Route of administration: IM injection
  Arms: Group 2 TIV-HA formulation 2 at high dose
Biological: RSV/hMPV/PIV3 formulation 2 at low dose — Suspension for injection in a vial. Route of administration: IM injection
  Arms: Group 8 RSV/hMPV/PIV3 formulation 2 at low dose
Biological: RSV/hMPV/PIV3 formulation 1 at high dose — Suspension for injection in a vial. Route of administration: IM injection
  Arms: Group 5 RSV/hMPV/PIV3 formulation 1 at high dose
Biological: RSV/hMPV/PIV3 formulation 2 at high dose — Suspension for injection in a vial. Route of administration: IM injection
  Arms: Group 6 RSV/hMPV/PIV3 formulation 2 at high dose
Biological: RSV/hMPV/PIV3 formulation 1 at low dose — Suspension for injection in a vial. Route of administration: IM injection
  Arms: Group 7 RSV/hMPV/PIV3 formulation 1 at low dose
Biological: RIV4 (Supemtek®) — Solution for injection in a prefilled syringe. Route of administration: IM injection
  Arms: Group 9 recombinant influenza vaccine quadrivalent (RIV4)

SUMMARY:
The objective of this study is to evaluate the safety and immunogenicity of different vaccines of hemagglutinin formulations of trivalent influenza vaccine or of a combined respiratory syncytial virus / human metapneumovirus / parainfluenza virus type 3 vaccine in healthy participants 18 to 49 years of age. A lipid nanoparticle will be used in this study.

Overall, the study is designed to:

* Assess the safety profile of the candidate formulations
* Describe the immunogenicity profile of the candidate formulations
* Eligible participants will be randomized to receive a single intramuscular injection of either one of the vaccine formulations.

Participants will be provided with a diary to solicit reporting of injection site reactions and systemic reactions, unsolicited Adverse Events (AEs), Serious Adverse Events (SAEs) and Adverse Events of Special Interest AESIs).

Participants will also be required to record their daily temperature on the diary.

DETAILED DESCRIPTION:
The duration of study participation will be approximately 6 months for each participant.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 49 years on the day of inclusion
* A female participant is eligible to participate if she is not pregnant or breastfeeding and one of the following conditions applies:

  * Is of non-childbearing potential. To be considered of non-childbearing potential, a female must be post-menopausal for at least 1 year, or surgically sterile OR
  * Is of childbearing potential and agrees to use an effective contraceptive method or abstinence from at least 4 weeks prior to study intervention administration until at least 4 weeks after study intervention administration.

Exclusion Criteria:

- Any medical condition or circumstance which, in the opinion of the investigator, might interfere with the evaluation of the study objectives

Note: The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 270 (Actual)
Dates: Start 2025-03-19 (Actual); Primary Completion 2025-12-11 (Actual); Study Completion 2025-12-11 (Actual)

PRIMARY OUTCOMES:
Presence of any unsolicited systemic Adverse Events (AEs) reported within 30 minutes after vaccination | Within 30 minutes after each vaccination
  Number of participants with unsolicited systemic AEs
Presence of solicited injection site and systemic reactions (ie, pre-listed in the participant's diary and in the eCRF (electronic case report form) occurring through 7 days after vaccination | Through 7 days after each vaccination
  Number of participants with solicited injection site and systemic reactions
Presence of unsolicited AEs reported through 28 days after vaccination | Through 28 days after each vaccination
  Number of participants with unsolicited AEs
Presence of SAEs (Serious Adverse Events) and AESIs (Adverse Events of Special Interest) throughout the study | Throughout study, approximately 6 months
  : Number of participants with SAEs and AESIs
Presence of out-of-range biological test results (including shift from baseline values) through 7 days after vaccination | Through 7 days after vaccination
  : Number of participants with out-of-range biological tests
Hemagglutinin Inhibition Assay (HAI) antibody (Ab) response to each homologous influenza strain at Day 1 and Day 29 | Day 1 and Day 29
RSV A, hMPV A and PIV3 serum neutralizing antibodies (nAb) titers at Day 1 and Day 29 | Day 1 and Day 29

SECONDARY OUTCOMES:
RSV B and hMPV A nAb titers at Day 1 and Day 29 | Day 1 and Day 29
Neutralization Test (NT) Ab response to each homologous influenza strain at Day 29 | Day 29

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (6):
- Australia (6):
  - Paratus Clinical, Blacktown, New South Wales
  - Paratus Clinical, Herston, Queensland
  - University of Sunshine Coast Clinical Trials, Morayfield, Queensland
  - University of Sunshine Coast Clinical Trials, South Brisbane, Queensland
  - Griffith University, Southport, Queensland
  - Emeritus Research, Camberwell, Victoria

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org